CLINICAL TRIAL: NCT05733507
Title: Efficacy of Simultaneous Infusion of Tirofiban With Intravenous Thrombolysis in Patients With Acute Anterior Choroidal Infarction or Paramedian Pontine Infarction
Brief Title: Tirofiban Plus Intravenous Thrombolysis in Acute Anterior Choroidal Infarction or Paramedian Pontine Infarction
Acronym: TITACIPPI
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Sud Francilien (Other)
Responsible Party: Sponsor
Other Study IDs: 2022/0039
Record Dates: First submitted 2023-02-08; First posted 2023-02-17 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Acute Anterior Choroidal Infarction (ACI); Paramedian Pontine Infarction (IPP)
Keywords: anterior choroidal infarction; paramedian pontine infarction; intravenous thrombolysis; tirofiban
MeSH Terms: interventions — Tenecteplase; Tissue Plasminogen Activator

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Intravenous thrombolysis (IVT): group of patients treated with IVT alone
  Interventions: Procedure: IVT with tenecteplase or alteplase
- Tirofiban + IVT: groups of patients treated with simultaneous infusion of tirofiban and IVT
  Interventions: Procedure: Intervention Name : Tirofiban and IVT with tenecteplase or alteplase

INTERVENTIONS:
Procedure: IVT with tenecteplase or alteplase — Patients received intravenous tenecteplase 0.25mg/kg (maximum dose: 25mg), administered as a bolus over 5 to 10 seconds or intravenous alteplase 0.9 mg/kg (maximum dose: 90mg), 10% as bolus and the remainder as continuous perfusion over 1 hour.
  Groups: Intravenous thrombolysis (IVT)
Procedure: Intervention Name : Tirofiban and IVT with tenecteplase or alteplase — IVT with tenecteplase or alteplase with continuous infusion of tirofiban 0.4µg/kg/min continued for 24 to 48 hours.
  Groups: Tirofiban + IVT

SUMMARY:
TITACIPPI (Tirofiban with Intravenous Thrombolysis in Acute Anterior Choroidal Infarction [ACI] and Paramedian Pontine Infarction [IPP]) study aimed to evaluate the efficacy and safety of simultaneous infusion of tirofiban with intravenous thrombolysis (IVT + tirofiban group) compared to IVT alone (IVT alone group) in patients with ACI or PPI. TITACIPPI study is a retrospective, single-center observational study conducted from March 01, 2014, to December 31, 2022.

DETAILED DESCRIPTION:
ACI and PPI are frequently associated with clinical fluctuations, characterized by recurrent transient more or less regressive stereotyped episodes of focal motor deficits affecting the face, arm, and leg, and finally with a risk of lasting neurological worsening that can lead to definite residual neurological disability. These ischemic strokes (ACI and PPI) are not very sensitive to IVT, thus 26% to 48% will experience neurological aggravation despite the administration of this treatment. Studies in Asia have shown a possible clinical benefit of simultaneous infusion of tirofiban with IVT in patients with ischemic stroke of atheromatous or microatheromatous origin without additional bleeding risk. To date, no studies have tested the efficacy of simultaneous infusion of tirofiban and IVT in the well-defined subgroup of ACI and PPI and a non-Asian population.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥ 18 years with ACI or PPI between March 01, 2014 and December 31, 2022.
* Patients hospitalized in the stroke unit of Centre Hospitalier Sud Francilien in the acute phase of their ischemic stroke (FLAIR negative on the pre-treatment brain MRI allowing IVT).
* Patients with NIHSS ≥ 2 on admission
* Patients treated with IVT
* For the experimental group: patients treated with tirofiban at 0.4 μg/kg/min with the start of infusion within 1 hour of IVT initiation.
* Patients with post-treatment brain MRI within 24-36h.

Exclusion Criteria:

* Patients with contraindications to IVT (cardiac, thoracic or digestive surgery less than 14 days old, thrombocytopenia < 100,000/mm3, etc.).
* Absence of MRI as initial imaging.
* Less than 24 hours of continuous infusion of tirofiban.
* Patients at high risk of cerebral hemorrhage: severe microangiopathy (Fazekas Score 3), microbleeds > 5, or leptomeningeal hemosiderosis suggestive of amyloid angiopathy.
* Patients with pre-stroke mRS ≥ 3.
* Patients informed of the research and objecting to the collection of their data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study included all patients aged ≥ 18 years with ACI or PPI, negative on FLAIR of the MRI of pretreatment, who had received IVT alone or simultaneous infusion of tirofiban with IVT in the stroke unit of CHSF between March 1, 2014, and December 31, 2022.
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2023-04-03 (Actual); Primary Completion 2023-09-13 (Actual); Study Completion 2023-09-13 (Actual)

PRIMARY OUTCOMES:
Volume of the ischemic lesion | at 24 hours
  Evolution of the volume of the ischemic lesion in diffusion-weighted imaging between initial MRI and post-therapy MRI

SECONDARY OUTCOMES:
NIHSS | at day 7
  NIHSS (from 0=favorable to 42=unfavorable)
Modified Rankin Scale (mRS) | at 3 months
  Proportion of the patients with mRS 0-2
Secondary neurological deterioration | at 72 hours
  Rate of secondary neurological deterioration (fluctuations or neurological progression defined as an increase of at least 1 point in NIHSS).
Cerebral hemorrhages | at 24 hours
  Rates of cerebral hemorrhages defined according to the Heidelberg Bleeding Classification
Systemic bleedings | at 24 hours
  Rate of significant systemic bleeding (i.e., requiring specific treatment).

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Sud Francilien, Corbeil-Essonnes, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Toudou-Daouda M, Soumah D, Bentamra L, Aminou-Tassiou NR, Baby M, Lhermitte Y, Altarcha T, Aghasaryan M, Smadja D, Chausson N. Efficacy of simultaneous infusion of tirofiban with intravenous thrombolysis in patients with acute anterior choroidal or paramedian pontine infarction: TITACIPPI study. Front Neurol. 2026 Jan 22;16:1692576. doi: 10.3389/fneur.2025.1692576. eCollection 2025. PMID 41659978